CLINICAL TRIAL: NCT03239392
Title: A Dose-Ranging Study of Intravenous BNZ132-1-40 in Patients With Large Granular Lymphocyte Leukemia or Refractory Cutaneous T-Cell Lymphoma
Brief Title: A Dose-Ranging Study of IV BNZ-1 in LGL Leukemia or Refractory CTCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bioniz Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNZ1-CT-201
Record Dates: First submitted 2017-07-31; First posted 2017-08-04 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2020-04

CONDITIONS: LGL Leukemia; CTCL
Keywords: BNZ-1; Cytokine; IL-2; IL-15
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BNZ-1 (Experimental): IV PEGylated BNZ132-1-40
  Interventions: Drug: BNZ132-1-40

INTERVENTIONS:
Drug: BNZ132-1-40 — Injectable PEGylated peptide antagonist that binds to the common gamma chain (γc) signaling receptor for the cytokines interleukin (IL)-2, IL-9, and IL-15
  Other Names: BNZ-1

SUMMARY:
This study is an open-label, multi-center, dose-ranging study to characterize the safety, tolerability, preliminary efficacy, and PK/PD of up to four dose levels of BNZ-1 administered weekly by IV infusion to adults diagnosed with Large Granular Lymphocyte (LGL) Leukemia or refractory Cutaneous T-cell Lymphoma (CTCL).

DETAILED DESCRIPTION:
This study is an open-label, multi-center, dose-ranging study to characterize the safety, tolerability, preliminary efficacy, and PK/PD of up to four dose levels of BNZ-1 administered weekly by IV infusion to adults diagnosed with LGL or CTCL. The study has 5 periods:

* Screening Period
* 4-week Treatment Period
* 3-month Treatment Extension Period
* Long-term Extension Period (open-ended)
* 6-week Follow-up Period Subjects will be screened for eligibility within 30 days of study Day 1 (first dosing day of the 4-Week Treatment Period).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to consent and participate in the study.
* Agrees not to receive any other investigational product or therapy while participating in this study.
* Must be:

  * Currently using two forms of effective birth control (one of which is a barrier method) for the duration of the study for both males and females of childbearing potential. Effective methods of birth control include hormonal contraception (i.e., birth control pills, injected hormones, vaginal ring), intrauterine device, or barrier methods with spermicide (i.e., diaphragm with spermicide, condom with spermicide), or
  * Surgically sterile (i.e., hysterectomy, tubal ligation, vasectomy).
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 to 2.
* Life expectancy >1 year.

LGL-Specific:

* Phenotypic studies (obtained within 8 weeks prior to study drug administration) from peripheral blood showing CD3+, CD57+ cells >400/mm³ or CD8+ cells >650/mm³.

  * Note: Complete blood count (CBC) and differential should be reported for the phenotyped sample.
* Evidence for clonal T-cell receptor gene rearrangement (obtained within 1 year prior to study drug administration).

CTCL-Specific:

* Histopathologically confirmed mycosis fungoides or Sézary syndrome (CTCL stage IIB or greater according to the European Organization for Research and Treatment of Cancer/International Society for Cutaneous Lymphomas [EORTC-ISCL] consensus classification) at study entry with progressive, persistent, or recurrent disease who have no available remaining standard therapeutic options (i.e., Refractory) as determined by the Investigator.

Exclusion Criteria:

* Clinically relevant hepatic, neurological, pulmonary, ophthalmological, endocrine, renal, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult, or that would put the subject at risk by participating in the study in the opinion of the Investigator.
* History of or currently active primary or secondary immunodeficiency.
* Known active bacterial, viral, fungal, mycobacterial infection, or other infection (including tuberculosis [TB] or atypical mycobacterial disease [but excluding fungal infection of nail beds, minor upper respiratory tract infection, and minor skin conditions]), or any major episode of infection that required hospitalization or treatment with IV antibiotics within 30 days of study drug administration or oral antibiotics within 14 days prior to study drug administration.
* Received other investigational products or therapy in the 60 days prior to study drug administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and relationship of treatment-emergent adverse events | 1 month
Incidence, severity and relationship of treatment-emergent adverse events | 4 months

SECONDARY OUTCOMES:
Pharmacodynamics | 16 weeks
  Flow cytometry: Change from baseline over time for Tregs, NK cells and CD8+ central memory T-cells
Single-dose and steady-state Cmax | 16 weeks
  Plasma levels of BNZ-1 will be measured after the 1st and last doses
Single-dose and steady-state AUC | 16 weeks
  Plasma levels of BNZ-1 will be measured after the 1st and last doses
Steady-state Elimination half-life (t1/2) | 16 weeks
  Plasma levels of BNZ-1 will be measured after the last dose

OTHER OUTCOMES:
Exploratory assessment of changes from baseline in CTCL disease severity (mSWAT) | 16 weeks
  mSWAT
Exploratory assessment of Complete Response in LGL | 16 weeks
  Normalization of CBC and LGL count
Exploratory assessment of Partial Response in LGL | 16 weeks
  ANC: >50% improvement from baseline and >500 cells/uL; or >50% reduction in transfusion requirements

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Brammer, MD, PhD, Principal Investigator — Ohio State University
Locations (4):
- United States (4):
  - City of Hope National Medical Center, Duarte, California
  - Moffitt Cancer Center, Tampa, Florida
  - The James Cancer Center, Ohio State University, Columbus, Ohio
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after study data analysis is completed and a CSR has been generated

REFERENCES:
- [Derived] Brammer JE, Ballen K, Sokol L, Querfeld C, Nakamura R, Mishra A, McLaughlin EM, Feith D, Azimi N, Waldmann TA, Tagaya Y, Loughran T. Effective treatment with the selective cytokine inhibitor BNZ-1 reveals the cytokine dependency of T-LGL leukemia. Blood. 2023 Oct 12;142(15):1271-1280. doi: 10.1182/blood.2022017643. PMID 37352612